CLINICAL TRIAL: NCT01394549
Title: Causes, Analysis of the Sub-evaluating Coronary Syndromes Acute and Disparities in France in Women
Acronym: CASSANDRE
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Stephane MANZO-SILBERMAN, Assistant Professor, French Cardiology Society
Other Study IDs: 11320
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Coronary Acute Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiology: The study includes all patients hospitalized for acute coronary syndrome during the week selected and who agreed to participate in the study.

SUMMARY:
Despite efforts of learned societies, community cardiology and more generally of most players in the health, cardiovascular diseases continue to be the leading cause of death among women in France and all over the Western world, there where they fell to second place among men. Clinical practice and the disparity between the sexes are still insufficiently known.

Multicenter observational study on a cross-week comparative basis with men

DETAILED DESCRIPTION:
In France, as in other industrialized countries, ischemic heart disease is a major cause of morbidity and mortality in women. Work to improve epidemiological knowledge, prevention, screening, risk stratification and treatment of ischemic heart disease in women has a potential impact on all the issues listed.

There is therefore a double challenge:

* A public health issue to alert the female population on cardiovascular risk and its consequences, while the female population does not feel concerned by the potential danger.
* A challenge for health professionals so that they have the same thing vis-à-vis the cardiovascular prevention among women and whatever their field of practice.

ELIGIBILITY:
Inclusion Criteria:

* Women all patients and / or men regardless of age
* Admitted to a cardiology department (in the intensive care unit or cardiology traditional) week of the survey,
* Having presented an acute coronary syndrome, regardless of the type with or without ST segment above, with or without elevated troponin, complicated or not, regardless of its support invasive or conservative,
* Patients who agreed to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in cardiac services regardless of the type of hospital where they are
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Clinical practices | 1 day
  To assess clinical practices and disparities between men and women in the management of acute coronary syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Background] WRITING GROUP MEMBERS; Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Roger VL, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):e46-e215. doi: 10.1161/CIRCULATIONAHA.109.192667. Epub 2009 Dec 17. No abstract available. PMID 20019324
- [Background] Stramba-Badiale M, Fox KM, Priori SG, Collins P, Daly C, Graham I, Jonsson B, Schenck-Gustafsson K, Tendera M. Cardiovascular diseases in women: a statement from the policy conference of the European Society of Cardiology. Eur Heart J. 2006 Apr;27(8):994-1005. doi: 10.1093/eurheartj/ehi819. Epub 2006 Mar 7. PMID 16522654
- [Background] Bairey Merz CN, Shaw LJ, Reis SE, Bittner V, Kelsey SF, Olson M, Johnson BD, Pepine CJ, Mankad S, Sharaf BL, Rogers WJ, Pohost GM, Lerman A, Quyyumi AA, Sopko G; WISE Investigators. Insights from the NHLBI-Sponsored Women's Ischemia Syndrome Evaluation (WISE) Study: Part II: gender differences in presentation, diagnosis, and outcome with regard to gender-based pathophysiology of atherosclerosis and macrovascular and microvascular coronary disease. J Am Coll Cardiol. 2006 Feb 7;47(3 Suppl):S21-9. doi: 10.1016/j.jacc.2004.12.084. PMID 16458167
- [Background] Lerner DJ, Kannel WB. Patterns of coronary heart disease morbidity and mortality in the sexes: a 26-year follow-up of the Framingham population. Am Heart J. 1986 Feb;111(2):383-90. doi: 10.1016/0002-8703(86)90155-9. PMID 3946178
- [Background] Michos ED, Nasir K, Braunstein JB, Rumberger JA, Budoff MJ, Post WS, Blumenthal RS. Framingham risk equation underestimates subclinical atherosclerosis risk in asymptomatic women. Atherosclerosis. 2006 Jan;184(1):201-6. doi: 10.1016/j.atherosclerosis.2005.04.004. PMID 15907856
- [Background] Kwok Y, Kim C, Grady D, Segal M, Redberg R. Meta-analysis of exercise testing to detect coronary artery disease in women. Am J Cardiol. 1999 Mar 1;83(5):660-6. doi: 10.1016/s0002-9149(98)00963-1. PMID 10080415
- [Background] Mieres JH, Shaw LJ, Arai A, Budoff MJ, Flamm SD, Hundley WG, Marwick TH, Mosca L, Patel AR, Quinones MA, Redberg RF, Taubert KA, Taylor AJ, Thomas GS, Wenger NK; Cardiac Imaging Committee, Council on Clinical Cardiology, and the Cardiovascular Imaging and Intervention Committee, Council on Cardiovascular Radiology and Intervention, American Heart Association. Role of noninvasive testing in the clinical evaluation of women with suspected coronary artery disease: Consensus statement from the Cardiac Imaging Committee, Council on Clinical Cardiology, and the Cardiovascular Imaging and Intervention Committee, Council on Cardiovascular Radiology and Intervention, American Heart Association. Circulation. 2005 Feb 8;111(5):682-96. doi: 10.1161/01.CIR.0000155233.67287.60. Epub 2005 Feb 1. PMID 15687114
- [Background] Einstein AJ, Moser KW, Thompson RC, Cerqueira MD, Henzlova MJ. Radiation dose to patients from cardiac diagnostic imaging. Circulation. 2007 Sep 11;116(11):1290-305. doi: 10.1161/CIRCULATIONAHA.107.688101. No abstract available. PMID 17846343
- [Background] Alexander KP, Chen AY, Roe MT, Newby LK, Gibson CM, Allen-LaPointe NM, Pollack C, Gibler WB, Ohman EM, Peterson ED; CRUSADE Investigators. Excess dosing of antiplatelet and antithrombin agents in the treatment of non-ST-segment elevation acute coronary syndromes. JAMA. 2005 Dec 28;294(24):3108-16. doi: 10.1001/jama.294.24.3108. PMID 16380591